CLINICAL TRIAL: NCT03007134
Title: Multicenter International Cross-Sectional Evaluation of Pulmonary Alveolar Proteinosis Trial
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-1204; RR019498 (Other Grant/Funding Number: NIH Office of Rare Disease Research)
Record Dates: First submitted 2016-11-28; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective Chart Review — No intervention.

SUMMARY:
The purpose of this study is to (1) compare a technically improved assay with an existing assay used to measure serum anti-GM-CSF antibodies in stored serum samples previously obtained from patients diagnosed with either primary, secondary, congenital or idiopathic pulmonary alveolar proteinosis (PAP), other chronic diseases or disease-free, healthy individuals; (2) determine the prevalence and levels of anti-GM-CSF autoantibodies and (3) define the breadth of the autoimmune antibody responses in primary PAP patients from the United States, Japan, Australia, and Europe using previously collected serum samples; and (4) using a chart review approach, compare the clinical, radiologic and laboratory features of primary PAP patients to determine if differences exist among patients in these globally geographically distributed regions.

DETAILED DESCRIPTION:
The Rare Lung Disease Consortium (RLDC), a group of geographically-dispersed clinical research sites, has been established to conduct collaborative clinical research regarding rare lung diseases. The collaborative work includes diagnostic, therapeutic and other studies in patients with pulmonary alveolar proteinosis (PAP), lymphangioleiomyomatosis (LAM), alpha-1 antitrypsin deficiency (AATD), or hereditary interstitial lung diseases. These patients can have delayed or incorrect diagnoses, and sub-optimal clinical management. The present protocol is focused to individuals with PAP.

PAP occurs as primary, secondary, congenital and idiopathic forms. RLDC investigators have previously shown that primary PAP is strongly associated with high levels of circulating, neutralizing anti-GM-CSF autoantibodies. Absence of GM-CSF bioactivity is thought to impair alveolar macrophage and blood neutrophil functions including reduced surfactant catabolism (alveolar macrophages - thought to result in surfactant accumulation in primary PAP) and immune dysfunction (neutrophil dysfunction, and possibly macrophage dysfunction - thought to increase the risk of infection in primary PAP). Secondary PAP is caused by an underlying condition believed to impair alveolar macrophage surfactant catabolism. Secondary PAP is related to other conditions, including myelogenous leukemias, infections and environmental exposures. Congenital PAP is caused by mutations in the genes encoding surfactant protein (SP)-B, SP-C or the ABCA3 transporter. Idiopathic PAP is that which results from unknown mechanisms. Anti-GM-CSF autoantibodies appear to be absent in secondary, congenital and idiopathic PAP.

This cross sectional study protocol is designed to evaluate the autoimmune aspect of PAP in patients that are currently being followed by clinical investigators in the Rare Lung Disease Consortium (RLDC). The study involves a retrospective chart review and serological analysis of preexisting, stored serum samples from individuals diagnosed with PAP. Thus, this study will not involve any direct interactions or contact with PAP patients or any other study participants. It will yield diagnostic information regarding the use of anti-granulocyte macrophage-colony stimulating factor (GM-CSF) autoantibody testing in patients with PAP. It will also yield information about the extent of the autoimmune response in primary PAP. In addition, the study will compare/contrast the clinical phenotypes of individuals with anti-GM-CSF autoantibody-positive PAP in various regions of the world. A stringent evaluation of the autoimmune aspects of PAP including rigorous anti-GM-CSF antibody testing will provide a better understanding of PAP and is expected to confirm the usefulness of serum anti-GM-CSF antibody testing in the clinical diagnosis of PAP. The study will evaluate the rate of serious or opportunistic infections and other clinical and demographic data from patients in various regions of the world to determine if significant differences exist, which will provide important knowledge regarding infectious and other complications associated with PAP.

ELIGIBILITY:
Inclusion Criteria:

Data and Serum must be from individuals of any age with confirmed diagnosis of PAP based on the following criteria:

* Radiographic features consistent with PAP
* Pathological or cytological findings consistent with PAP determined by either open lung biopsy, transbronchial biopsy or bronchoalveolar lavage cell/fluid cytology.
* Elevated anti-GM-CSF autoantibody concentration, when available

Ability of the international PI's and their research coordinators to ship samples in compliance with this study.

Exclusion Criteria:

* No established diagnosis of PAP
* Incomplete chart records in which >25% of the requested data is unable to be confirmed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Autoimmune PAP
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Standardize the anti-GM-CSF autoantibody ELISA | 1 year
  To compare a novel assay to an existing assay used to measure anti-GM-CSF autoantibodies in banked serum samples previously collected from individuals diagnosed with primary, secondary, congenital or idiopathic PAP, other chronic disorders, or disease-free, healthy individuals.

SECONDARY OUTCOMES:
Geographic distribution of anti-GM-CSF autoantibody levels | 1 years
  GM-CSF autoantibody concentration in patients with autoimmune PAP
Breadth of the autoimmune antibody phenotype of individuals with autoimmune PAP | 3 years
  Autoimmune antibody phenotype of individuals with autoimmune PAP
Age of onset PAP symptoms | 2 years
  Range of age at onset of symptoms of PAP among PAP patients from different global geographic regions
Age at the time of definitive PAP diagnosis | 2 years
  Range of age at the time of definitive pathologic diagnosis of PAP among PAP patients from different global geographic regions
Length of time from onset of symptoms and definitive diagnosis of autoimmune PAP | 2 years
  Length of time between the onset of symptoms and a definitive pathologic diagnosis of PAP among PAP patients from different global geographic regions
Gender distribution among PAP patients | 2 years
  Gender distribution among PAP patients from different global geographic regions
Tobacco use among PAP patients | 2 years
  Variability of tobacco use among PAP patients from different global geographic regions
Major medical history comparison among PAP patients | 2 years
  Variability of associated major medical diagnoses among PAP patients from different global geographic regions
Disease severity variability among autoimmune PAP patients from various geographic locations | 2 years
  Severity of the disease at onset among PAP patients from different global geographic regions
Number of secondary infections that occur in patients with primary PAP | 2 years
  Number of participants documented to have had a secondary infection(s)
Type of secondary infections that occur in patients with primary PAP | 2 years
  List the specific organisms documented to have infected PAP patients

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (6):
- United States (2):
  - Brody School of Medicine, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Ruhrlandklinik Essen, Essen, Germany
- Clinica Malattie Apparato Respiratorio Università di Pavia, Pavia, Italy
- Japan (2):
  - University of Niigata Medical and Dental School, Niigata
  - NHO Kinki-Chuo Chest Center, Osaka

IPD SHARING:
Plan to Share IPD: No